CLINICAL TRIAL: NCT02716727
Title: Comparison of Two Gingival Displacement Procedures; a Randomized Clinical Trial
Brief Title: Comparison of Two Gingival Displacement Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-1787
Record Dates: First submitted 2016-03-10; First posted 2016-03-23 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-07

CONDITIONS: Gingival Retraction Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aquasil Ultra Cordless, Dentsply (Active Comparator): Gingival displacement procedure that uses a pneumatic hand piece to inject the light body impression material into the gingival sulcus.
  Interventions: Device: Aquasil Ultra Cordless, Dentsply
- Ultrapak, Ultradent cord (Active Comparator): The knitted cord is used for physical displacement of gingival tissue. Cord is placed in the gingival sulcus and left in place for at least 4 minutes to achieve gingival displacement.
  Interventions: Device: Ultrapak, Ultradent cord

INTERVENTIONS:
Device: Aquasil Ultra Cordless, Dentsply — Cordless gingival displacement procedure
  Arms: Aquasil Ultra Cordless, Dentsply
Device: Ultrapak, Ultradent cord — Cordless gingival displacement procedure
  Arms: Ultrapak, Ultradent cord

SUMMARY:
Purpose: To compare the quality of impressions made with a cordless gingival displacement procedure versus impressions made with a corded technique. The devices and materials used in both procedures are FDA-approved, marketed, and will be used according to label.

Participants: Approximately sixty (60) adult patients who are treatment planned for indirect restorations (crowns) at the UNC School of Dentistry. Procedures (methods): Participants will be randomized to receive either the cordless gingival displacement procedure (Aquasil Ultra Cordless, Dentsply), or the corded technique (Ultrapak, Intradent) followed by impression with Aquasil Ultra, Dentsply. Participants will complete the Faces pain scale. Impressions will be photographed, digitally scanned, and evaluated.

DETAILED DESCRIPTION:
Background: Indirect fixed prosthodontic restorations are widely used for the restoration of teeth. The fabrication of a well-fitting indirect restoration requires an accurate impression which captures the cervical finish line. Dentists have a hard time making proper impressions, with a reported 56% of impressions sent to labs being inadequate. The most common deficiency is inadequate recording of the cervical finish line. The primary reason for this inadequacy is deficient gingival displacement technique. More effective and efficient gingival displacement procedure can lead to clinically improved fixed restorations, less patient chair time, and less patient discomfort.

Materials and Methods: Sixty (60) patients will be recruited from the University of North Carolina (UNC) School of Dentistry (SOD), and they will be randomly split into 2 equal sized groups: 30 patients cordless gingival displacement procedure (Aquasil Ultra Cordless, Dentsply International); 30 patients traditional corded technique using Aquasil Ultra Polyvinyl siloxane (PVS) impression material, Dentsply International, gingival displacement cord (Ultrapak, Ultradent Products International) hydrated with aluminum chloride hexahydrate (Hemodent, Premier Dental Products Company). Patient inclusion criteria include: 1) requires indirect restoration/s. 2) probing depths 4mm or less. 3) No bleeding on probing. 4) finish line 0-1mm sub-gingival.

Specific Aims:

1. To examine if a cordless gingival displacement procedure can properly displace gingival tissue to facilitate acceptable impressions that accurately capture the prepared cervical finish line for the fabrication of indirect fixed prosthodontic restorations. These impressions will be digitally scanned, and then all of the impression scans will be evaluated for acceptability based on a set of criteria (evaluation form). The evaluations will be conducted by 2 standardized individuals.
2. To determine if a cordless gingival displacement procedure facilitates impressions that area at least as good as the traditional corded gingival displacement procedure. The impression scans will be evaluated and then a comparison will be made between the 2 groups of impressions.
3. To determine if a cordless gingival displacement procedure is more time efficient than the traditional corded procedure. All procedures will be timed, starting when the gingival displacement procedure is commenced and ending when the impression is removed from the patient's mouth.
4. To determine if a cordless gingival displacement procedure causes less trauma and discomfort to the patient than the traditional corded procedure. Patient discomfort will be evaluated with a 3 question written survey (0-10 scale answers).

The hypothesis contemplated in this proposal explores if a cordless gingival displacement procedure can properly displace gingival tissues to facilitate an acceptable impression that accurately captures the prepared cervical finish line for the fabrication of indirect fixed prosthodontic restorations. Our objective is to identify if a new procedure can improve the efficiency of a traditionally technique-sensitive procedure in dentistry.

Materials and Methods:

A total of sixty participants will be recruited from the University of North Carolina (UNC) School of Dentistry (SOD) Graduate Prosthodontics clinic, Graduate Operative clinic, and the Dental Faculty Practice. There will be two (2) randomly assigned groups; thirty (30) patients who will receive a cordless gingival displacement procedure (Aquasil Ultra Cordless, Dentsply International) and thirty (30) patients who will receive the traditional gingival displacement technique with retraction cord (UltraPak, Ultradent Products International) hydrated with aluminum chloride hexahydrate (Hemodent, Premier Dental Products Company), and impression made with Polyvinyl siloxane (PVS) impression material (Aquasil Ultra, Dentsply International).

Any indirect restoration requires an accurate impression of the prepared margins and the tooth. To obtain an accurate impression, the gingiva has to be displaced or retracted temporarily to allow for the impression material to flow into the gingival sulcus and capture the margins of the preparation. Traditionally this is accomplished by packing two knitted cords. The cordless technique does not require this step but uses a pneumatic hand piece through which the light body impression material is injected in the sulcus displacing the gingival tissue in order to capture the margins of the prepared tooth. Both techniques are described in detail below.

Traditional Corded Impression Procedure:

1. The prepared tooth is rinsed and dried, and assure hemostasis.
2. Small diameter retraction cord, after it has been hydrated with Hemodent (hemostatic agent) for 10 minutes, is tucked around the tooth in the space between it and its surrounding gum tissue. A second larger diameter retraction cord, also hydrated with Hemodent, will be placed over the first cord and tucked around the tooth. These cords will be left in place for a minimum of 8 minutes. These cords temporarily push the gum tissue away from the tooth.
3. After a minimum of 8 minutes, the larger 2nd cord will be removed, and the tooth dried. Quickly, after confirmation of a dry field, the light body consistence impression material is dispensed using a plastic syringe around the prepared tooth and across the occlusal surfaces of adjacent teeth.
4. An impression tray that has been filled with the heavy body consistency impression material is then placed over the arch of teeth, and gently pressed into place to ensure the teeth are completely covered with a uniform thickness of impression material. As the different impression material consistencies set, they fuse together into a single unit.
5. When removed from the mouth, the impression should contain a negative copy of both the prepared tooth and the teeth of that jaw.

Cordless Impression Procedure:

1. The prepared tooth is rinsed and dried, and assure hemostasis.
2. Apply B4 + surface optimizer (manufacturer recommended for increasing the wettability of the prepared tooth).
3. Using the digit power dispenser (pneumatic hand piece that connects to the dental chair), unit dose cartridge, and intrasulcular plastic mixing tip, depress foot pedal and gently insert the plastic tip into the gingival sulcus of the prepared tooth, slightly apical to the preparation finish line. Material should flow into the gingival sulcus making sure to have impression material ahead of the intrasulcular tip as you move around the tooth and the prepared finish line.
4. An impression tray that has been filled with the heavy body consistency impression material is then placed over the arch of teeth, and gently pressed into place to ensure the teeth are completely covered with a uniform thickness of impression material. As the different impression material consistencies set, they fuse together into a single unit.
5. When removed from the mouth, the impression should contain a negative copy of both the prepared tooth and the teeth of that jaw.

Post Impression:

Once the impressions are made, the clinician will record the type of impression material used; whether tray adhesive was used; the tray material; the type of tray used; and the number of units requested. The impressions will be photographed and digitally scanned and then collectively evaluated at a later time, based on a criteria evaluation form by two calibrated evaluators. The evaluator will assess each impression for errors in the finish line; in the tray/material; and errors with gingival displacement/hemostasis as primary outcomes. The number of errors can range from 0 to 13.

Two secondary outcomes will also be analyzed. First, the time required to perform the impression procedure will be recorded using a timer. Second, patient discomfort will be assessed using the FACES visual picture pain scale rated from 1-10 based on the following question posed at 3 points during treatment; "How much discomfort are you experiencing at this point in treatment?" This question will be asked before the impression procedure is initiated, immediately after the impression procedure is completed, and again at the completion of the treatment appointment. Each question will be rated on a scale of 1 to 10. The total score indicated by the sum of the 3 questions will be analyzed.

As part of this study, the participant might be seen one or two times, one for consenting to participate in the study and another time for treatment and impression; we may be able to complete both during the same appointment. The consent appointment will ideally occur simultaneously with their consultation/treatment planning appointment prior to treatment.

The proposed research study will approximately include a total of 60 participants. Recruitment of the patient population will rely on referrals from UNC School of Dentistry (UNC SOD) Faculty Practice, UNC SOD dental student's clinic (DDS student clinics, graduate student clinics and DFP). Apart from participating in the study, the patient may seek other dental treatments in the above mentioned clinics.

Study clinicians will be calibrated on both the cordless and the corded gingival displacement procedures and impression procedures in a practice session. Clinical instruction protocols will be printed on laminated forms for all study clinicians to follow, for both the cordless and the corded procedures. These clinical protocol forms will be in the clinicians operatory during actual study treatment, and this protocol must be followed for the impression to be included in the study.

On the day of the appointment, participants will be requested to sign a consent form. The study subject will be asked to complete the standard adult medical and dental health history questionnaire provided by the UNC SOD and will be provided with the UNC Chapel Hill Notice of Privacy Practices and the Consent for Purposes of Treatment, payment and health care operation. Other than the screening consent, these are standard practices followed by UNC SOD for all patients. The study is mandated to adhere to theses protocols prior to treating a patient at the UNC SOD. An oral examination will be performed by the research dentist to evaluate if the patient meets inclusion criteria, after the subject has signed all documents. Upon consent to participate, appointments will be made for treatment at UNC SOD, as it would happen as part of their regular treatment.

Second appointment - during this scheduled time, a clinical re-evaluation will be completed, and if appropriate, treatment will be completed. Clinical data will be collected prior to starting the treatment; we will collect soft tissue response [Bleeding on Probing (BoP) and Probing Pocket Depth (PPD)]. Customary anesthesia and tooth preparation will be performed by the clinician as necessary for the particular indirect restoration, and when completed, the finish line will be evaluated for inclusion criteria by the clinician. If all inclusion criteria are met, a coin toss will determine which gingival displacement procedure will be performed, and the gingival displacement procedure and impression will be made as described in this study protocol and as followed on the laminated clinical protocol sheet. If the clinician finds that the first impression is inadequate and chooses to make an additional impression, only the first impression will be evaluated for the study and a note will be indicated to record the number of impressions the clinician made to achieve an acceptable impression. If the inclusion criteria are not met, a clinically appropriate impression method will be performed at the clinician's judgment and will be made per case by the treating clinician, following standard of care for the treatment that the patient receives.

Patients will be given appropriate verbal and written post-procedure instructions; and appointments will be made for restoration try-in and delivery, as would happen as part of their regular treatment. There are no potential direct benefits to the participant besides the fact that particularly close attention will be paid to the gingival displacement and impression procedures, and there will be close evaluation of impressions.

All of the impressions will be photographed and digitally scanned, and also given a number which will be recorded on a master sheet with the type of gingival displacement procedure indicated. No other patient identifiers will be included. These scans will be evaluated collectively on a later day, and will be critiqued based on a criteria form. This evaluation will be performed by 2 investigators, and will be completed independently. Impressions will be deemed acceptable or not acceptable, and the reasons for not acceptable impressions will be indicated. The evaluation criteria are listed in Appendix B.

The scientific knowledge to be gained will be the efficacy of a new gingival displacement procedure, and if it can be adopted to improve patient treatment and treatment outcomes. The risks of the study are consistent with the current standard of care. Standard treatment protocols will be observed for the treatment of teeth which require indirect restorations. The risks will be minimized by treatment evaluation and proper treatment technique.

Data monitoring Research data management will involve collection, entry, processing, storage, retrieval, archival, distribution and documentation of information. Data collection will adhere to precise written forms. Data will be stored in a series of Microsoft Access data files, which will be accessible to the Investigators and their staff. Only project-related personnel will be able to access these files. Data collection forms will be kept in locked files. Quality assurance (QA) will occur as data is entered in order to check for data completeness and consistency prior to entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be adult males or females over the age of 18.
* Patients must be able and willing to follow study procedures and instructions.
* Patients must have read, understood and signed an informed consent form.
* Patients must be in good general health.
* Patient must require one or more indirect restorations.
* Probing pocket depths around the treatment tooth/teeth must be 4mm or less.
* There must be no bleeding on probing around the treatment tooth/teeth.
* The prepared finish line must be between 0 to 1mm sub-gingival (inclusive).

Exclusion Criteria:

* Individuals who have a chronic disease with oral manifestations.
* Individuals who exhibit gross oral pathology.
* Smokers, Diabetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumitha Ahmed, BDS, MS, Principal Investigator — UNC-Chapel Hill
Locations (1):
- UNC School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (15.01) | 65.0 (9.03) | 60.5 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Errors in Impressions Made for Indirect Restorations
Description: Impressions will be assessed for technique errors
Time Frame: Through impression completion, an average of 10-20 minutes or when impression material is completely set
Measure: Number; unit: percentage of impressions
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord
Number analyzed (Participants) | 7 | 9
percentage of impressions
  Voids/Bubbles | 85.7 | 33.3
  Lack of Wash Material | 28.6 | 44.4
  Tearing | 71.4 | 11.1
  Cotton Roll Attached | 0 | 11.1
  Inadequate Fusion Between Wash & Tray Material | 57.1 | 11.1
  Lack of Polymerization | 14.3 | 0
  Inadequate Retention | 0 | 0
  Pressure of Tray on Soft Tissue | 0 | 11.1
  Void on Preparation | 85.7 | 88.8
  Show-through of Occlusal/Incisal Edges | 0 | 22.2
  Tissue Over Finish Line | 42.9 | 11.1
  Retraction Cord Attached | 0 | 11.1
  Blood on the Impression | 0 | 33.3

2. Primary Outcome: Mean Time Required to Make the Impression
Description: The time required to perform the impression procedures from the start of the gingival displacement procedure to completion of impression.
Time Frame: Through impression completion, an average of 10-20 minutes or when impression material is completely set
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord
Number analyzed (Participants) | 7 | 9
minutes | 5.92 (8.57) | 9.81 (8.57)

3. Primary Outcome: Mean Patient Discomfort Scores
Description: Patient discomfort will be assessed using the Wong-Baker FACES Pain Rating Scale™.The FACES Pain Scale is a dimensionless 10-point Likert scale used to assess self-reported pain intensity on a scale from 0 (no pain) to 10 (most pain you can imagine). Greater pain scores are indicative of more severe pain. Patients self-reported pain using the FACES evaluation at the beginning of the appointment, immediately before start of impression procedure, immediately after the impression procedure completed, and at the end of the appointment.
Time Frame: From start of visit until the end of the visit, approximately 3 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord
Number analyzed (Participants) | 7 | 9
score on a scale
  Start of Visit | 7.64 (6.03) | 8.31 (6.03)
  Immediately Before Starting Impression | 8.64 (7.87) | 7.43 (7.87)
  Immediately After Impression Completed | 1.85 (1.57) | 2.12 (1.45)
  At End of Visit | 8.00 (7.58) | 8.00 (7.58)

4. Secondary Outcome: Comparison of Percentage of Impression Errors Made by Residents and Faculty
Description: Accuracy of the impression assessed for technique errors based on the clinical experience of the provider.
Time Frame: Through impression completion, an average of 10-20 minutes or when impression material is completely set
Population: Due to loss of key study personnel these data were not collected.
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Comparison of the Time Required to Make Impressions Between Residents and Faculty
Description: The time required to perform the impression procedures from the start of the gingival displacement procedure to completion of impression based on the clinical experience of the provider.
Time Frame: Through impression completion, an average of 10-20 minutes or when impression material is completely set
Population: Due to loss of key study personnel these data were not collected.
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mean Patient Discomfort Score Comparison for Procedures Completed by Residents and Faculty
Description: Patient discomfort will be assessed based on the clinical experience of the provider using the Wong-Baker FACES Pain Rating Scale™.The FACES Pain Scale is a dimensionless 10-point Likert scale used to assess self-reported pain intensity on a scale from 0 (no pain) to 10 (most pain you can imagine). Greater pain scores are indicative of more severe pain. Patients self-reported pain using the FACES evaluation at the beginning of the appointment, immediately before start of impression procedure, immediately after the impression procedure completed, and at the end of the appointment.
Time Frame: From start of visit until the end of the visit, approximately 3 hours
Population: Due to loss of key study personnel these data were not collected.
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Comparison of Percentage of Impression Errors Based on Maxillary and Mandibular Arch
Description: Accuracy of the impression assessed for technique errors based on the location of the tooth in the mouth (maxillary and mandibular arch).
Time Frame: Through impression completion, an average of 10-20 minutes or when impression material is completely set
Population: Due to loss of key study personnel these data were not collected.
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Comparison of the Time Required to Make Impressions in the Maxillary and Mandibular Arch
Description: The time required to perform the impression procedures from the start of the gingival displacement procedure to completion of impression based on the location of the tooth in the mouth (maxillary and mandibular arch).
Time Frame: Through impression completion, an average of 10-20 minutes or when impression material is completely set
Population: Due to loss of key study personnel these data were not collected.
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Mean Patient Discomfort Score Comparison Based on Maxillary and Mandibular Arch
Description: Patient discomfort will be assessed based on the location of the tooth in the mouth (maxillary and mandibular arch) using the Wong-Baker FACES Pain Rating Scale™.The FACES Pain Scale is a dimensionless 10-point Likert scale used to assess self-reported pain intensity on a scale from 0 (no pain) to 10 (most pain you can imagine). Greater pain scores are indicative of more severe pain. Patients self-reported pain using the FACES evaluation at the beginning of the appointment, immediately before start of impression procedure, immediately after the impression procedure completed, and at the end of the appointment.
Time Frame: Through impression completion,an average of 10-20 minutes or when impression material is completely set
Population: Due to loss of key study personnel these data were not collected.
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of signing Informed Consent until participant left the clinic following completion of procedure, a total of approximately 3 hours.
Arm/Group | Aquasil Ultra Cordless, Dentsply | Ultrapak, Ultradent Cord
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT02716727/Prot_SAP_000.pdf